CLINICAL TRIAL: NCT04024618
Title: A Pilot Feasibility Study of Nutritional Outcomes in Autologous Hematopoietic Stem Cell Transplant Recipients Comparing Enteral Nutrition Versus Parenteral Nutrition
Brief Title: Feasibility Study Comparing Enteral vs Parenteral Nutritional Outcomes in Autologous Stem Cell Transplant Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LHSC BMT19.01
Record Dates: First submitted 2019-04-24; First posted 2019-07-18 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2019-07

CONDITIONS: Malignant Hematologic Neoplasm
Keywords: Non- Hodgkin's Lymphoma; Hodgkin's Lymphoma; Multiple Myeloma; AHSCT
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma | interventions — Parenteral Nutrition; Enteral Nutrition

STUDY DESIGN:
Intervention Model Description: Randomization will be 1:1, both EN and PN arms. The patients will be randomized in permutated blocks independently by Statistician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parenteral Nutrition (Active Comparator): Patients who have been randomized to receive PN will be started on day 5 post AHSCT. This will be if patient intake is < 80% of usual oral intake at that time. The central venous catheter required for PN administration will be already in place for AHSCT treatment, prior to admission and pre-transplant evaluation. Nutritional support will continue until oral intake is >50% or until the patient is ready for discharge if intake remains < 50% of recommendations.
  Interventions: Procedure: Parenteral Nutrition/Enteral Nutrition
- Enteral Nutrition (Experimental): Patients who have been randomized to receive EN will have a Nasogastric tube (NGT) inserted on day 5 post AHSCT, prior to start of Enteral feeds. This would be a polyurethane tube, 8-10 French, which will be inserted by physician or Nurse Practitioner with position confirmed by radiological examination. This will be if patient intake is < 80% of usual oral intake at that time. Nutritional support will continue until oral intake is >50% or until the patient is ready for discharge if intake remains < 50% of recommendations.
  Interventions: Procedure: Parenteral Nutrition/Enteral Nutrition

INTERVENTIONS:
Procedure: Parenteral Nutrition/Enteral Nutrition — Patients randomized to the parenteral nutrition arm will receive nutrition by IV and patients randomized to the enteral nutrition arm will receive nutrition by NG tube.

SUMMARY:
This study will highlight that Enteral Nutrition (EN) is as effective in nutritionally supporting as Parenteral Nutrition (PN) in this group of patients undergoing an autologous hematopoietic stem cell transplantation (AHSCT). The rationale of this study is to compare nutritional, medical, cost and Quality of Life (QOL) outcomes in patients receiving either EN or PN nutritional support in patients. The main outcomes are to examine are nutritional status, medical complications, cost and QOL before and after AHSCT.

DETAILED DESCRIPTION:
This will be a pilot open randomized study. The study will be conducted at the inpatient setting at London Health Sciences Centre in London, ON. Forty patients will be randomized in permutated blocks independently by Statistician, to either the EN or PN group on admission to the unit. The baseline evaluations are blood work, Bioelectric Impedance Analysis (BIA), Subjective Global Assessment (SGA), Body Mass Index (BMI) calculation, ultrasound, and a medical evaluation. Patients do have the right to refuse either or both types of nutritional support. As part of standard care, the risks and benefits of nutritional support for both EN and PN will be explained to the patient.

Consent will be obtained prior to admission. Most of these patients initially continue to maintain their oral intake even after chemotherapy. On Day 5+/- 1 day after transplantation, the randomized nutrition therapy will only be initiated only if patient intake is < 80% of usual intake, where they will be provided with 25-35 kcal/kg/day, 1.2-1.5g of protein/kg/day, and omega-3 to supplement any oral intake the patient might not have. If the intake is >80% of required intake, initiation of randomized therapy will only happen on the day the intake falls to <80% of required nutritional intake.

Patients will be monitored until Day 15 where post-transplant evaluations will be conducted: blood work, BIA, SGA, ultrasound, BMI, food records, and medical evaluation. If at that time, patients are not consuming 50% of energy from oral feeds, nutrition therapy will continue until oral goal is met or until discharge for medical reasons. Patients will be assessed at Day+30 post-transplant in clinic and the following will be completed blood work, BIA, SGA, BMI, food records, ultrasound, medical complications and a QOL assessment.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients aged 18 to 75 years.
* Patients admitted to Victoria Hospital undergoing AHSCT on C7 unit.
* Patient consented to participate in the study
* Patients diagnosed with the following conditions: Non- Hodgkin's Lymphoma (all types), Hodgkin's Lymphoma (all subtypes) and Multiple Myeloma
* Patients receiving any of the following: Conditioning chemotherapy: Melphalan, Etoposide/Melphalan, or Carmustine, Etoposide, Cytarabine, Melphalan
* Have a functional Gastrointestinal tract

Exclusion Criteria:

* Intestinal obstruction
* Patients with nasal deformities, tumors of nasal tracts or upper nare obstruction.
* Patients with active bacteremia while proceeding with transplant
* Patients with active malignancy of Upper GI tract, not in remission as evidenced by recent imaging studies (< 4 weeks)
* Patients with any GI bleeding, paralytic ileus, obstruction, or any other GI condition which excludes use of the GI system for nutritional support as these patients will require PN feeding only and cannot be randomized

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Enrollment of patients | 30 days
  The number of patients enrolled

SECONDARY OUTCOMES:
quadriceps muscle layer thickness | 21 days
  Maintenance and/or improvement of quadriceps muscle layer thickness (QMLT) measurement: measured by ultrasound.
Duration of Support | 21 days
  A comparison of duration in days a patient will require enteral or parenteral nutritional support during their admission.
Changes in costs | 21 days
  The cost of daily total PN is $80/day and cost of EN feeds would be $40/day. This is a 50% change in costs.
Hospital Stay | 21 days
  Length of hospital stay (decrease by 1+/-2 days)
Mortality | 30 days
  Mortality on Day+30 Post AHSCT
Changes in body fat | 21 Days
  Measuring the changes in percentage of body fat mass using Bioelectric Impedance Analysis
Changes in Lean Muscle | 21 Days
  Measuring the changes in percentage lean muscle mass using Bioelectric Impedance Analysis
Changes in costs to hospital when using enteral nutritional | 21 Days
  the measurement the length of their stay in the hospital by days, fewer days of hospitalization = lower costs and more days of hospitalization = greater costs
Transition from EN to oral feeding | 15 Days
  Successful transition from EN to oral feeding versus Parenteral Nutrition to oral feeding defined by 50% oral intake on Day+15 of AHSCT.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre-Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan on sharing individual participant data to other researchers

REFERENCES:
- [Background] Sekine L, Ziegelmann PK, Manica D, da Fonte Pithan C, Sosnoski M, Morais VD, Falcetta FS, Ribeiro MR, Salazar AP, Ribeiro RA. Frontline treatment for transplant-eligible multiple myeloma: A 6474 patients network meta-analysis. Hematol Oncol. 2019 Feb;37(1):62-74. doi: 10.1002/hon.2552. Epub 2018 Sep 20. PMID 30129104
- [Background] Gisselbrecht C, Van Den Neste E. How I manage patients with relapsed/refractory diffuse large B cell lymphoma. Br J Haematol. 2018 Sep;182(5):633-643. doi: 10.1111/bjh.15412. Epub 2018 May 29. PMID 29808921
- [Background] Lipkin AC, Lenssen P, Dickson BJ. Nutrition issues in hematopoietic stem cell transplantation: state of the art. Nutr Clin Pract. 2005 Aug;20(4):423-39. doi: 10.1177/0115426505020004423. PMID 16207682
- [Background] Buono R, Longo VD. Starvation, Stress Resistance, and Cancer. Trends Endocrinol Metab. 2018 Apr;29(4):271-280. doi: 10.1016/j.tem.2018.01.008. Epub 2018 Feb 17. PMID 29463451
- [Background] Deeg HJ, Seidel K, Bruemmer B, Pepe MS, Appelbaum FR. Impact of patient weight on non-relapse mortality after marrow transplantation. Bone Marrow Transplant. 1995 Mar;15(3):461-8. PMID 7599573
- [Background] August DA, Huhmann MB; American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.) Board of Directors. A.S.P.E.N. clinical guidelines: nutrition support therapy during adult anticancer treatment and in hematopoietic cell transplantation. JPEN J Parenter Enteral Nutr. 2009 Sep-Oct;33(5):472-500. doi: 10.1177/0148607109341804. No abstract available. PMID 19713551
- [Background] Roberts S, Miller J, Pineiro L, Jennings L. Total parenteral nutrition vs oral diet in autologous hematopoietic cell transplant recipients. Bone Marrow Transplant. 2003 Oct;32(7):715-21. doi: 10.1038/sj.bmt.1704204. PMID 13130320
- [Background] Bozzetti F, Braga M, Gianotti L, Gavazzi C, Mariani L. Postoperative enteral versus parenteral nutrition in malnourished patients with gastrointestinal cancer: a randomised multicentre trial. Lancet. 2001 Nov 3;358(9292):1487-92. doi: 10.1016/S0140-6736(01)06578-3. PMID 11705560
- [Background] Seguy D, Berthon C, Micol JB, Darre S, Dalle JH, Neuville S, Bauters F, Jouet JP, Yakoub-Agha I. Enteral feeding and early outcomes of patients undergoing allogeneic stem cell transplantation following myeloablative conditioning. Transplantation. 2006 Sep 27;82(6):835-9. doi: 10.1097/01.tp.0000229419.73428.ff. PMID 17006332
- [Background] Lach K, Peterson SJ. Nutrition Support for Critically Ill Patients With Cancer. Nutr Clin Pract. 2017 Oct;32(5):578-586. doi: 10.1177/0884533617712488. Epub 2017 Jun 20. PMID 28633000
- [Background] Seguy D, Duhamel A, Rejeb MB, Gomez E, Buhl ND, Bruno B, Cortot A, Yakoub-Agha I. Better outcome of patients undergoing enteral tube feeding after myeloablative conditioning for allogeneic stem cell transplantation. Transplantation. 2012 Aug 15;94(3):287-94. doi: 10.1097/TP.0b013e3182558f60. PMID 22785249
- [Background] Zhang G, Zhang K, Cui W, Hong Y, Zhang Z. The effect of enteral versus parenteral nutrition for critically ill patients: A systematic review and meta-analysis. J Clin Anesth. 2018 Dec;51:62-92. doi: 10.1016/j.jclinane.2018.08.008. Epub 2018 Aug 8. PMID 30098572
- [Background] Beckerson J, Szydlo RM, Hickson M, Mactier CE, Innes AJ, Gabriel IH, Palanicawandar R, Kanfer EJ, Macdonald DH, Milojkovic D, Rahemtulla A, Chaidos A, Karadimitris A, Olavarria E, Apperley JF, Pavlu J. Impact of route and adequacy of nutritional intake on outcomes of allogeneic haematopoietic cell transplantation for haematologic malignancies. Clin Nutr. 2019 Apr;38(2):738-744. doi: 10.1016/j.clnu.2018.03.008. Epub 2018 Mar 28. PMID 29650256
- [Background] Kiss N, Seymour JF, Prince HM, Dutu G. Challenges and outcomes of a randomized study of early nutrition support during autologous stem-cell transplantation. Curr Oncol. 2014 Apr;21(2):e334-9. doi: 10.3747/co.21.1820. PMID 24764716
- [Background] Barbosa-Silva MC, Barros AJ, Wang J, Heymsfield SB, Pierson RN Jr. Bioelectrical impedance analysis: population reference values for phase angle by age and sex. Am J Clin Nutr. 2005 Jul;82(1):49-52. doi: 10.1093/ajcn.82.1.49. PMID 16002799
- [Background] Tillquist M, Kutsogiannis DJ, Wischmeyer PE, Kummerlen C, Leung R, Stollery D, Karvellas CJ, Preiser JC, Bird N, Kozar R, Heyland DK. Bedside ultrasound is a practical and reliable measurement tool for assessing quadriceps muscle layer thickness. JPEN J Parenter Enteral Nutr. 2014 Sep;38(7):886-90. doi: 10.1177/0148607113501327. Epub 2013 Aug 26. PMID 23980134